CLINICAL TRIAL: NCT01633099
Title: The Clinical Research About the Therapeutic Effect and Safety of 10 Days Regimen With Single-agent of Decitabine for Elderly AML Patients
Brief Title: Therapeutic Effect and Safety Study of Decitabine in Elderly Acute Myeloid Leukemia Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jianxiang Wang (Unknown)
Collaborators: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jianxiang Wang, deputy director, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DACOGENAML2003
Record Dates: First submitted 2012-06-24; First posted 2012-07-04 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Untreated Adult Acute Myeloid Leukemia; Effect of Drugs; Drug Safety
Keywords: decitabine; acute myeloid leukemia; elderly patient
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine, CR rate,OS,EFS,RFS (Other): Therapeutic effect and safety of 10 days of decitabine. Acute myeloid leukemia,no acute promyelocytic leukemia.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — 1. Number of Cycles: 4 cycles.
  2. Dose and drug delivery(decitabine):
  The 1st cycle: 20 mg/m2, (iv,>1 hour) d1-10 of each 28 day cycle. The 2nd-4th cycle:If bone marrow blast cells≥5%, the following cycle is the same as the 1st cycle.
  If bone marrow blast cells<5%, the following cycle:decitabine 20 mg/m2, (iv,>1h) on d1-5 of each 28 day cycle.
  If Grade 4 neutropenia（<0.5×10E9/L）come arise after 5 days' cycle of decitabine and lasts more than 14 days in last cycle,the next cycle will decrease dose to 4 days(20 mg/m2, IV ,>1h, on d1-4 of each 28 day cycle).If Grade 4 neutropenia（<0.5×10E9/L）come arise after 4 days' cycle of decitabine and lasts more than 14 days in last cycle,the next cycle will decrease dose to 3 days(20 mg/m2, IV,>1h, on d1-3 of each 28day cycle).
  Other Names: Dacogen

SUMMARY:
The purpose of this study is to confirm the safety and the therapeutic effect of Decitabine in the treatment of elderly Acute Myeloid Leukemia (AML) patients.

DETAILED DESCRIPTION:
The outcome of the elderly AML patients is very poor. No obvious progress was achieved in this field. Decitabine is a kind of specific DNA methylation shift enzyme inhibitor. It can reverse the DNA methylation and induce the differentiation and apoptosis of the tumor cells. Recent studies about decitabine in the treatment for elderly AML patients had achieved inspiring results and indicated that low dose decitabine maybe a good choice for elderly AML patients. So in this research the investigators plan to evaluate the safety and the therapeutic effect of decitabine in the treatment of elderly AML patients.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of acute myeloid leukemia.De novo or secondary AML.
2. Age >= 60years,female and male.
3. Before the enrollment，WBC < 40×10E9/L，Plt > 20×10E9/L（Hydroxyurea is permitted.）
4. In 2 weeks before the enrollment，total bilirubin < 1.5×ULN，ALT < 2.5×ULN；GGT < 2.5×ULN ，Scr < 2.0×ULN or creatinine clearance rate ≥ 50 ml/min（Cockroft-Gault）.
5. Before the enrollment，patients must be free from the toxicity caused by the former treatment.Received no chemotherapy in the last 4 weeks and no nitrosourea in the last 6 weeks.
6. Contraception must be taken to avoid pregnancy during the study.
7. ECOG 0,1, or 2, predicted lifetime longer than 12 weeks.
8. Patients must sign the informed consent prior to any study related screening procedures being performed.

Exclusion Criteria:

1. Acute promyelocytic leukemia.
2. Chromosome and genetic abnormalities related with t（8; 21）、inv（16）、t（15; 17）.
3. Central nervous system leukemia.
4. Bone marrow dry tap.
5. Patients received stem cell transplantation or chemotherapy containing azacitidine,cytarabine or decitabine in last one year, radiation therapy in last 14 days,lenalidomide in 30 days before included.
6. Patients suffered from autoimmune hemolytic anemia or immune thrombocytopenia.
7. Patients suffered from non-leukemia related comorbidities that will cause dysfunction of organs.
8. Patients suffered from unstable angina or （NYHA）3/4 Congestive heart failure.
9. Patients suffered from chronic respiratory disease and needed continued oxygen.
10. Other active malignancy.
11. Active HBV,HCV or AIDS patients.
12. Uncontrolled virus or bacterium infection.
13. The investigator believe that patients who are not suitable for this trial.
14. Severe mental or body disorders which will interfere the research such as uncontrolled heart,lung diseases,diabetes,etc.
15. Allergic to decitabine or its accessory.
16. Patients received other researches in last 30 days.
17. Without contraception.
18. Complications causing organ dysfunction which are not caused by AML.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Complete response rate after induction chemotherapy with decitabine | 21 days after the induction chemotherapy
Overall survival rate | Up to 46 months after inclusion
Event free survival rate | Up to 46 months after inclusion
Relapse free survival rate | Up to 46 months after inclusion

SECONDARY OUTCOMES:
Adverse events of decitabine for elderly AML patients | Up to 46 months
Weight of elderly AML patients | Up to 46 months
ECOG(Eastern Cooperative Oncology Group) score for elderly AML patients | Up to 46 months
Physical examination of decitabine for elderly AML patients | Up to 46 months
Blood pressure of elderly AML patients | Up to 46 months
Respiratory rate of elderly AML patients | Up to 46 months
Heart rate of elderly AML patients | Up to 46 months
Body temperature of elderly AML patients | Up to 46 months
ECG of elderly AML patients | Up to 46 months
Bone marrow condition of elderly AML patients | Up to 46 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, MD, Principal Investigator — Institute of Hematology, Hospital of Blood Disease, Chinese Academy of Medical Sciences

REFERENCES:
- [Background] Burnett AK, Milligan D, Prentice AG, Goldstone AH, McMullin MF, Hills RK, Wheatley K. A comparison of low-dose cytarabine and hydroxyurea with or without all-trans retinoic acid for acute myeloid leukemia and high-risk myelodysplastic syndrome in patients not considered fit for intensive treatment. Cancer. 2007 Mar 15;109(6):1114-24. doi: 10.1002/cncr.22496. PMID 17315155
- See also: We do not have a protocol's home page. This website is our hospital's home page and introduces some information of our hospital. — http://www.chinablood.com.cn/